CLINICAL TRIAL: NCT04893044
Title: Alcohol Misuse Intervention in Active Duty US Navy Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: New York University (Other); John Jay College of Criminal Justice, City University of New York (Other)
Responsible Party: Principal Investigator, Braden Hale, Faculty, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 190366
Record Dates: First submitted 2021-04-27; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Alcohol Drinking; Alcohol Use Disorder
Keywords: Military
MeSH Terms: conditions — Alcohol Drinking; Alcoholism | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: Randomized pilot trial of video intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure (Experimental): These participants watched a 3 minute long video prior to a long weekend. The intent was to see if watching the video altered their alcohol consumption compared to a group that did not watch the video. Urine alcohol metabolites were measured before and after the weekend.
  Interventions: Behavioral: Video
- Control (No Intervention): These participants did not watch a video, and their urine alcohol metabolites were measures at the same dates as the exposure group above.

INTERVENTIONS:
Behavioral: Video — The video was a 3 minutes and based on "inoculation theory" to modify behavior towards moderating the effect of alcohol use as opposed to advising no use at all.
  Arms: Exposure

SUMMARY:
A pilot trial among ship-board US Navy personnel surrounding a holiday weekend tested an evidence-based video on responsible drinking.

Service members >18 years were eligible to volunteer if they were aboard during data collection. Participants were randomized to intervention or control arms, with all given a brief survey before (T1) and after (T2) the weekend. The intervention arm viewed a 3-minute video at T1. A urine specimen collected at T1 and T2 for ethyl glucuronide (EtG) measurement used >100ng/ml for significant alcohol use. Multivariable regression measured odds of detecting EtG at T2, controlling for T1 EtG detectability, age, and alcohol misuse at baseline per AUDIT-C.

86 subjects participated at T1, and 100 at T2, with complete data for 72 (control, n=34; intervention, n=38) who participated in both T1 and T2 were analyzed. Average age was 28 years with 25% and 32% reporting white or black/African-American, 54% married and 84% <E6. At T1, 22% (n=16) and T2, 32% (n=23) had EtG>100ng/ml. At T1, 50% and 55% in control and intervention arms respectively, screened positive for alcohol misuse by AUDIT-C; T1 AUDIT-C screen positivity was significantly associated with detecting EtG>100ng/ml at T1 (p=0.04). Control arm EtG>100ng/ml participants increased 1.7-fold over the weekend, from n=7 at T1 to n=12 at T2; the intervention arm had no increase in EtG>100ng/ml participants, with n=11 at T1 and n=11 at T2.

DETAILED DESCRIPTION:
U.S. Navy active duty personnel were recruited to participate in a randomized pilot trial evaluating the efficacy of a 3 minute video intervention designed to promote safer drinking and reduce adverse consequences of alcohol use. All subjects were provided informed consent prior to participation. An incentive of a $5 gift card was provided upon completion of T1, and a $10 gift card provided after completion of T2. Subject participation and data were anonymous; personal identifiers were collected in order to link samples and surveys between timepoint 1 (T1) and timepoint 2 (T2), but after the linking, all identifier data were destroyed. To minimize risk associated with collecting personal identifiers, we did not retain any personal identifiers, to include sex categorization of participants. Subjects completed the T1 survey with only study ID on the form and were then asked to provide a urine sample.

Urine samples were collected in toilet facilities onboard the ship. The collections were not monitored. Urine samples were labelled with the subject ID number and stored at 4 degrees C until they could be shipped. For T1, samples remained refrigerated over the weekend as receiving personnel would not be available during the weekend; at T2, the samples were shipped the following day.

At T1, after providing the urine sample, the intervention subjects watched a 3 minute video, while the control subjects left the area without watching the video.

After the long weekend, subjects were asked to return to the study area, complete a brief survey, and provide a second urine specimen.

The 3 minute video was created for this pilot study. One of the authors with experience in inoculation theory (RJD) guided the content of the video, which was produced, directed and filmed at the New York University Film School.

The T1 surveys collected data on year of birth (as a verification in linking T1 and T2 data in event of linking error), demographic information to include race, relationship status, and pay grade. Additional questions included "have you ever had a drinking problem?", the AUDIT-C questions , and questions regarding if conflicts, accidents or other issues had occurred as a result of alcohol use.

The T2 survey collected year of birth (see above), AUDIT-C questions (modified to reflect data only from the preceding weekend), and the same questions regarding conflicts, accidents or other issues as a result of alcohol use.

Procedure for EtG testing Chemicals and materials Standards of ethyl glucuronide (EtG) and ethyl glucuronide-d5 (EtG-d5) were purchased at concentrations of 1 mg/mL in 1 mL methanol from Cerilliant Corp (Round Rock, TX, US). Liquid chromatography-mass spectrometry (LC-MS) grade methanol, acetonitrile and formic acid, and Sarstedt Inc 10 mL sc tubes 16x100 mm were purchased from Thermo Fisher Scientific (Waltham, MA, US). Nano-Filter vials ® 0.2 µm PES with pre-slit gray cap were from Thomson Instrument Company (Oceanside, CA, US).

Sample preparation: dilution and filtration One hundred µL of urine sample, 300 µL of water and 100 µL of the internal standard EtG-d5 at 0.5 µg/mL were vortex-mixed in a clean Starstedt tube. Two hundred µL of the sample were transferred into the shell vial of the Filter Vial. The plunger with filter was inserted all the way into the shell vial. Twenty µL of the filtered sample were directly injected into the LC-MS/MS.

Calibrators were prepared at concentrations 0.05, 0.1, 0.25, 0.5, 1, 5 and 10 µg/mL, and quality controls at 0.15 and 7.5 µg/mL, using 100 µL of blank urine, 200 µL of water, 100 µL of the corresponding working solution and 100 µL of the internal standard solution.

Instrumental analysis The chromatographic separation was carried out on a Nexera UHPLC system (Shimadzu, Columbia, MD, US). The Nexera UHPLC system consisted of two binary LC-20AD XR high-performance liquid chromatography pumps, online degassing unit (DGU-20A 3R), cooled autosampler (SIL-20A XR) and an oven (CTO-20AC). The column was a Hypercarb column (2.1x 100 mm, 3 µm) from Thermo Fisher Scientific. The mobile phase, 0.1 % formic acid in water (A) and acetonitrile (B), was delivered at a flow rate of 0.3 mL/min. Column temperature was 30C. The gradient began with B at 5% then increasing to 95% in 6 min. B at 95% was held for 0.5 min after which it decreased to 5%, and it was held for 1 min. Total run time was 7.5 min.

The mass spectrometer was a triple quadrupole LCMS-8050 from Shimadzu equipped with electrospray ionization source (ESI). The heating gas and drying gas flows were 15 and 10 L/min, respectively, with a nebulizing gas flow at 2 L/min. The interface temperature was 300°C and the heat block temperature was 400°C. All compounds were analyzed using ESI in negative ionization mode, and two transitions in multiple reaction monitoring (MRM) mode were acquired for each analyte.

Statistical analysis Statistical analyses were performed using Stata version 15.1 (StataCorp, College Station, TX). Descriptive statistics were calculated to characterize participant demographics and by alcohol use at T1 and T2. Fisher's exact tests were used for categorical variables with n<15 in any category and Wilcoxon rank-sum tests for non-normally distributed continuous variables to examine bivariate associations between the groups. All tests were two-sided with significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All members of selected US Navy ship are eligible

Exclusion Criteria:

* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Urinary ethyl glucuronide (EtG) | 3 days
  Alcohol metabolite

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test - Consumption (AUDIT-C) score | 3 days
  Measurement of self-reported alcohol consumption. The AUDIT-C score is scored on a scale from 0-12. The higher the AUDIT-C score is, the more likely it is to indicate a alcohol use disorder. In males, a score of 4 or higher is a positive screen. In women, a score of 3 or higher represents a positive screen. In this trial, we did not collect male/female data and used a cutoff of 4 for all participants.

CONTACTS AND LOCATIONS:
Locations (1):
- US Navy, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McDonell MG, Skalisky J, Leickly E, McPherson S, Battalio S, Nepom JR, Srebnik D, Roll J, Ries RK. Using ethyl glucuronide in urine to detect light and heavy drinking in alcohol dependent outpatients. Drug Alcohol Depend. 2015 Dec 1;157:184-7. doi: 10.1016/j.drugalcdep.2015.10.004. Epub 2015 Oct 9. PMID 26475403